CLINICAL TRIAL: NCT03985072
Title: Phase 1 Open-label Two-stage Safety and Tolerability Study With Subcutaneous Administration of Andes-1537 for Injection in Patients With Specific Types of Advanced Solid Tumors That Are Refractory To or No Available Standard Therapy
Brief Title: Study With Andes-1537 in Patients With Specific Types of Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andes Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB1537-002
Record Dates: First submitted 2019-05-17; First posted 2019-06-13 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Tumor, Solid; Gall Bladder Cancer; Cervical Cancer; Gastric Cancer; Pancreatic Cancer; Colorectal Cancer
Keywords: Neoplasm; Solid Tumor; Cancer; Carcinoma
MeSH Terms: conditions — Neoplasms; Gallbladder Neoplasms; Uterine Cervical Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Andes-1537 (Experimental): There will be 5 different cohorts each representing a different type of solid cancer (gallbladder and biliary tract cancer, cervical cancer, gastric cancer, pancreatic cancer, and colorectal cancer). All patients will receive a dose of 400 mg of Andes-1537 five days per week for continuous cycles of 4 weeks that will be repeated until the patients presents drug toxicity requiring treatment discontinuation or disease progression without any noted clinical benefit as assessed by the investigator.
  Interventions: Drug: Andes-1537 for Injection

INTERVENTIONS:
Drug: Andes-1537 for Injection — Andes-1537 administered subcutaneously five days per week.

SUMMARY:
The study is a Phase 1 Open-label Two-stage, Safety and Tolerability Study with Cancer Type-specific Cohorts, Evaluating Subcutaneous Administration of Andes-1537 for Injection in Patients with Advanced Solid Tumors that are Refractory to Standard Therapy or For Which No Standard Therapy Is Available. Patients with unresectable solid tumors that are refractory or have failed standard therapy and are deemed non-eligible or intolerant to further therapy or for which no standard therapy is available will be included in 5 cancer type-specific parallel cohorts. The following tumor types will be evaluated for potential inclusion in each cancer type-specific cohort: gallbladder & biliary tract carcinoma; cervical carcinoma; gastric carcinoma; pancreatic carcinoma, and colorectal carcinoma.

DETAILED DESCRIPTION:
After screening, 9 patients in each cancer type-specific cohort (gallbladder & biliary tract carcinoma; cervical carcinoma; gastric carcinoma; pancreatic carcinoma, and colorectal carcinoma) will enter stage 1. These patients will receive a dose of 400 mg of Andes-1537 five times per week for continuous cycles of 4 weeks that will be repeated until the patients presents drug toxicity requiring treatment discontinuation or disease progression with no noted clinical benefit as assessed by the investigator. The safety and tolerability evaluation will be continuous during the study. The efficacy evaluation will be done by analysis of the clinical objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria after patients complete the first two cycles (8 weeks). Thereafter, clinical ORR will be assessed every 8 weeks. Additionally, tumor-cell activity assessment will be performed in biopsy samples after the patients complete the first 2 cycles (8 weeks). Tumor markers assessment according to the type of tumor will be evaluated every 2 cycles and at the end of study (EOS) visit. Analysis of the tumor metabolic activity through the PET-CT scan and quality of life of patients through questionnaire will be evaluated every 2 cycles. As predefined and according with the decision of the Study Safety and Steering Committee (SSC), in those cohorts where minimal clinical response criteria were met or according to the decision of the SSC based on the risk / benefit analysis, considering toxicity criteria and observed biological responses, 15 additional patients will be recruited (total of 24 patients per cohort) for stage 2 of the study. Patients included in stage 2 will receive the same treatment regimen described for stage 1 and will be followed until the patients present disease progression or drug toxicity requiring treatment discontinuation. Patients included in stage 2 will receive the same follow-up as patients in stage 1.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years of age or older.
2. Can understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessment or procedure, and are able to adhere to the study visit schedule and other protocol requirements.
3. Patients with documented pathological evidence of advanced unresectable solid tumors that are, in the opinion of their treating physician, refractory or have failed standard therapy and are deemed non-eligible or intolerant to further therapy, or for which no standard therapy is available will be enrolled in both stages of the study in the following 4 cancer type-specific cohorts:

   * Gallbladder & Biliary Tract Cancer: Histologically confirmed stage 4 or unresectable stage 3b biliary tract & gallbladder adenocarcinoma with relapsed, refractory or progressive disease, who cannot tolerate or is considered resistant to platinum based chemotherapy for advanced disease such as cis-platinum and gemcitabine.
   * Cervical Cancer: Histologically confirmed stages 4 or 3b cervical cancer with relapsed, refractory or progressive disease, who cannot tolerate or is considered resistant to platinum based chemotherapy for advanced disease such as cis-platinum/carboplatin and paclitaxel.
   * Gastric Cancer: Histologically confirmed stage 4 or recurrent gastric adenocarcinoma with relapsed, refractory or progressive disease, who cannot tolerate or has progressed after first and second line combined chemotherapy regimens containing Epirubicin, cisplatin, fluorouracil (5-FU)/ leucovorin, oxaliplatin, irinotecan and/or docetaxel. Patients with Her2Neu positive cancer will not be eligible.
   * Pancreatic Cancer: Histologically confirmed stage 4 or recurrent pancreatic adenocarcinoma with relapsed, refractory or progressive disease, who cannot tolerate or is considered resistant to combined treatment with leucovorin calcium, 5-FU, irinotecan and oxaliplatin (FOLFIRINOX) or Gemcitabine based chemotherapy, depending on age and performance status.
   * Colorectal Cancer: Histologically confirmed Stage IV colorectal adenocarcinoma with relapsed, refractory, or progressive disease, who cannot tolerate or is considered resistant to combined treatment with fluoropyrimidines and/or oxaliplatin and/or irinotecan and/or Epidermal Growth Factor-1 (EGF1) inhibitors (depending on molecular profile) either as single agent or in combination therapy, depending treating oncologist´s decision. Patients with Kirsten rat sarcoma viral oncogene homolog (KRAS) - Neuroblastoma RAS Viral Oncogene Homolog (NRAS) wild type should have progressed after cetuximab or panitunumab unless contraindicated or not available.
4. Have measurable disease by RECIST.
5. Have Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 1.
6. Have life expectancy ≥ 12 weeks as judged by the investigator.
7. Have adequate organ function, confirmed by the following laboratory values obtained ≤ 3 days prior to the first treatment:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   * Hemoglobin (Hgb) ≥ 9 g/dL
   * Platelets ≥ 100 × 109/L
   * Aspartate aminotransaminase (AST) and alanine aminotransaminase (ALT) ≥ 2.5 × upper limit of normal (ULN)
   * Serum total bilirubin ≤ 2.0 × ULN
   * Serum creatinine ≤ 1.5 × ULN (patients with Creatinine > 1,5 x ULN may be considered to participate if estimated or measured creatinine clearance ≥ 60 mL/min)
   * Prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤ 1.5 ULN if not on anticoagulation therapy (patients receiving anticoagulation therapy must be in the therapeutic range and stable for ≥ 4 weeks prior to study entry)
8. Patients with accessible tumor tissue, susceptible to biopsies through procedures such as colonoscopy, endoscopy, endocervical biopsy (among others), are required to provide consent for two biopsies throughout the study, to analyze tumor biomarkers. The first tumor biopsy will be performed in these patients in a timeframe of 28 days prior to the initial administration of the investigational product Andes-1537. Alternatively, pathological archived material may be used, if the biopsy was collected within a period of two months prior to initiation of treatment and with no anti-cancer treatment performed since the collection date. The second biopsy will be performed after 2 cycles (8 weeks) of treatment. If no archival material is available, and only one lesion is amenable for biopsy (and is the only target lesion), the Medical Monitor should be consulted for subject eligibility. Tumor biopsies and tumor archival material must be suitable for biomarker assessment as described in the Laboratory Manual.
9. Female patients of childbearing potential must have a negative serum pregnancy test and be using adequate contraception (defined below) prior to study entry and must agree to continue to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Note: Options for adequate contraception with a failure rate of <1% per year include: tubal ligation, male sterilization, hormonal implants, established proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and cervical cap) may be combined to achieve a failure rate of <1% per year. Barrier methods must always be supplemented with the use of a spermicide. Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal or postovulation methods) and withdrawal are not acceptable methods of contraception. Should a female patient or a female partner of a male patient become pregnant or suspect she is pregnant while participating in the study or within 6 months following discontinuation of the study drug, the patient should inform the investigator immediately.

Exclusion Criteria:

1. Have known central nervous system metastases.
2. Have unstable angina, clinically significant cardiac arrhythmia, New York Heart Association Class 3 or 4 congestive heart failure, or prolonged QT interval corrected (QTc) wave of greater than 470 ms.
3. Receiving treatment with any medication known to produce QT prolongation within 7 days of study entry.
4. Have had prior systemic chemotherapy treatments or investigational modalities ≤ 5 half-lives (t1/2) or 4 weeks, whichever is shorter, prior to starting treatment with Andes 1537 or who have not recovered from side effects, grade 2 or greater, of such therapy (except alopecia).
5. Have had major surgery ≤ 2 weeks prior to starting treatment with Andes-1537 or who have not recovered from side effects of such surgery.
6. Are pregnant or breastfeeding.
7. Have had deep vein thrombosis (DVT) or venous thromboembolism within 6 weeks of study entry. Patients are permitted to enter the study if they are receiving anticoagulation therapy considered to be in the therapeutic range and are stable for ≥ 4 weeks prior to study entry.
8. Have active uncontrolled bleeding or a known bleeding disorder.
9. Have any serious or unstable concomitant systemic conditions that are incompatible with this clinical study, including but not limited to substance abuse, psychiatric disturbance, or uncontrolled intercurrent illness (including active infection), arterial thrombosis, or symptomatic pulmonary embolism.
10. Have a known sensitivity to any of the components of Andes-1537.
11. Are unable or unwilling to follow protocol instructions and requirements.
12. Have received more than 2 previous lines of systemic antineoplastic treatment that includes chemotherapeutic agents, target therapies, or immunotherapy considered as standard treatments for the type of tumor that the patient has.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) through stages 1 and 2 of the study | Screening and during cycle treatment (each cycle 4 weeks) until study completion (approximately 24 weeks or earlier if patient discontinues from study)
  Assessment of safety and tolerability through the incidence and severity of TEAEs from change in baseline for reported adverse events, safety labs, vital signs, electrocardiograms, and injection site reactions

SECONDARY OUTCOMES:
Objective response rate (ORR) according to RECIST | Assessment performed every 8 weeks following completion of 2 treatment cycles (each cycle 4 weeks) from screening to study completion until confirmed disease progression or Andes-1537 toxicity (approximately 24 weeks or earlier if patient discontinues)
  Computed tomography (CT) or magnetic resonance imaging (MRI) scan of tumors located in chest, abdomen, and pelvis every 8 weeks for change in tumor size from baseline measurements
Duration of response and duration of stable disease according to RECIST | Assessment performed every 8 weeks following completion of 2 treatment cycles (each cycle 4 weeks) from screening to study completion until confirmed disease progression or Andes-1537 toxicity (approximately 24 weeks or earlier if patient discontinues)
  CT or MRI of tumor every 8 weeks and compared to previous RECIST assessment
Progression free survival time according to RECIST | Assessment performed every 8 weeks following completion of 2 treatment cycles (each cycle 4 weeks) from screening to study completion until confirmed disease progression or Andes-1537 toxicity (approximately 24 weeks or earlier if patient discontinues)
  CT or MRI of tumor every 8 weeks and compared to previous RECIST assessment
Andes-1537 tumor-cell biomarker activity in biopsy tissue | Screening to end of cycle 2 (each cycle 4 weeks) treatment (approximately 8 weeks)
  Biopsies will be performed at screening prior to treatment and at the end of the second cycle of treatment in tumor tissue that is accessible by procedures such as colonoscopy, endoscopy, endocervical biopsy, etc. Tumor biopsy samples will be assessed for biomarkers of Andes-1537 activity through histology assays.
Plasma concentration of Andes-1537 after subcutaneous administration for pharmacokinetic (PK) parameter area under the plasma concentration versus time (AUC) | Screening and during cycle treatment (each cycle 4 weeks) until study completion (approximately 24 weeks or earlier if patient discontinues from study)
  Plasma samples will be collected in each treatment cycle for evaluation of AUC
Plasma concentration of Andes-1537 after subcutaneous administration for PK parameter maximum plasma concentration (Cmax) | Screening and during cycle treatment (each cycle 4 weeks) until study completion (approximately 24 weeks or earlier if patient discontinues from study)
  Plasma samples will be collected in each treatment cycle for evaluation of Cmax
Plasma concentration of Andes-1537 after subcutaneous administration for PK parameter time to maximum concentration (Tmax) | Screening and during cycle treatment (each cycle 4 weeks) until study completion (approximately 24 weeks or earlier if patient discontinues from study)
  Plasma samples will be collected in each treatment cycle for evaluation of Tmax
Plasma concentration of Andes-1537 after subcutaneous administration for PK parameter half-life (t1/2) | Screening and during cycle treatment (each cycle 4 weeks) until study completion (approximately 24 weeks or earlier if patient discontinues from study)
  Plasma samples will be collected in each treatment cycle for evaluation of t1/2
Incidence of Andes-1537 anti-drug antibodies (ADAs) in the plasma | Screening and during cycle treatment (each cycle 4 weeks) until study completion (approximately 24 weeks or earlier if patient discontinues from study)
  Assessment of immunogenicity of Andes-1537 following subcutaneous administration by determining the presence of Andes-1537 ADAs in all patients receiving at least 2 treatment cycles. Blood samples will be collected and stored for future analysis of ADAs prior to the first injection of cycle 1 and then every 8 weeks following completion of a treatment cycle, prior to beginning the next cycle, and end-of-study visit.

OTHER OUTCOMES:
Evaluate exploratory response of patient quality of life assessment | Assessment performed every 8 weeks following completion of 2 treatment cycles (each cycle 4 weeks) from screening to study completion until confirmed disease progression or Andes-1537 toxicity (approximately 24 weeks or earlier if patient discontinues)
  Patients to complete quality of life questionnaire
Evaluate the exploratory tumor response of metabolic activity | Assessment performed every 8 weeks following completion of 2 treatment cycles (each cycle 4 weeks) from screening to study completion until confirmed disease progression or Andes-1537 toxicity (approximately 24 weeks or earlier if patient discontinues)
  Tumor metabolic activity determined by positron emission tomography (PET) plus CT
Evaluate the exploratory response of inflammatory markers | Screening and during cycle treatment (each cycle 4 weeks) until study completion (approximately 24 weeks or earlier if patient discontinues from study)
  Change in plasma concentration from baseline of markers of inflammation for C-reactive protein and complement activity will be evaluated during the first cycle, every 2 weeks. After the first cycle, checked once per month following completion of a treatment cycle and prior to beginning the next cycle.
Evaluate the exploratory response of tumor markers | Assessment performed every 8 weeks following completion of 2 treatment cycles (each cycle 4 weeks) from screening to study completion until confirmed disease progression or Andes-1537 toxicity (approximately 24 weeks or earlier if patient discontinues)
  Change in plasma concentration of tumor markers cancer antigen (CA) 19-9 in biliary tract cancer and pancreatic carcinoma and carcinoembryonic antigen (CEA) tumor marker in colorectal carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadita Mendez, PhD, Study Director — Andes Biotechnologies
Locations (4):
- Chile (4):
  - Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan
  - Centro de Cancer de Nuestra Senora de la Esperanza, Red de Salud UC CHRISTUS, Santiago, Santiago Metropolitan
  - Instituto Nacional del Cáncer (INCANCER), Santiago, Santiago Metropolitan
  - Centro de Investigaciones Clinicas Vina del Mar, Viña del Mar, V Region de Valparaiso

IPD SHARING:
Plan to Share IPD: No